CLINICAL TRIAL: NCT01276600
Title: Dose-Proportionality and Intra-Individual Variability of Intracellular Tenofovir Diphosphate and Emtricitabine Triphosphate In Healthy Volunteers
Brief Title: Dose-Proportionality and Intra-Individual Variability of Intracellular TFV-DP and FTC-TP in Healthy Volunteers
Acronym: HPTN066
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HPTN 066
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HIV
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): 1 tablet orally weekly
  Interventions: Drug: Emtricitabine/tenofovir
- Arm 2 (Experimental): One tablet orally twice weekly
  Interventions: Drug: Emtricitabine/tenofovir
- Arm 3 (Experimental): Two tablets orally twice weekly
  Interventions: Drug: Emtricitabine/tenofovir
- Arm 4 (Experimental): One tablet orally daily
  Interventions: Drug: Emtricitabine/tenofovir

INTERVENTIONS:
Drug: Emtricitabine/tenofovir — 200mg of emtricitabine 300mg of tenofovir

SUMMARY:
Describe the dose-proportionality and intra-individual variability of tenofovir diphosphate (TFV-DP) and emtricitabine triphosphate (FTC-TP) at steady-state in healthy human participants taking Truvada® (FTC 200mg/TDF 300 mg) under direct observation.

DETAILED DESCRIPTION:
This PK study is designed to establish the dose-proportionality of TFV and FTC (serum and intracellular forms) with daily to weekly dosing. This information is essential to (1) employ drug concentration as an adherence measure in future PrEP studies, and (2) to estimate the anticipated concentration of parent and active moieties of TFV and FTC in intermittent PrEP regimens associated with full adherence to a prescribed regimen. In addition, intra-individual variability will be assessed to improve sample size estimates in future PrEP studies that use drug concentration as an adherence measure or where PK-PD correlations are planned. The dose-proportionality of intra-cellular phosphates of the two components of the study product has not previously been established. Given the complexity of movement of these drugs between body compartments (central compartment, vaginal mucosal tissue, vaginal lumen, gastrointestinal mucosal tissue, gastrointestinal lumen), into cells within these compartments, and intra-cellular phosphorylation, it is possible that non-dose proportional kinetics, such as mixed or zero-order saturable processes may be operating.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible for inclusion in this study:

* 18 to 44 years of age, inclusive on the date of screening.
* Provides informed consent for the study.
* Non-reactive HIV rapid test results at the screening and enrollment visits.
* An estimated calculated creatinine clearance (eCcr) at least 70 mL/min by the Cockcroft-Gault formula where:

  * eCcr (female) in mL/min = [(140 - age in years) x (weight in kg) x 0.85] / (72 x serum creatinine in mg/dL).
  * eCcr (male) in mL/min = [(140 - age in years) x (weight in kg)] / (72 x serum creatinine in mg/dL).
* Participants are sexually active, defined as at least one sex (vaginal or anal intercourse) act in the 30 days prior to screening.
* Participants must agree to use condoms for all coital events during study participation.
* Intensive sampling cohort only:

  * Not using spermicide as a means of birth control (in conjunction with a condom or diaphragm)
* Women must:

  * Be pre-menopausal
  * Have regular menstrual cycles with at least 21 days between menses (unless on contraception that causes amenorrhea or irregular menses)
  * Have a negative urine pregnancy test at screening and enrollment
  * Be utilizing an alternative method of birth control in addition to condoms (hormonal contraceptive, diaphragm or have undergone surgical sterilization) or have a vasectomized exclusive male partner.
  * Intensive sampling cohort only:

    * Have a cervix
    * Have documentation of a normal Pap smear within 12 months

Exclusion Criteria:

* At screening::

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 1.5 X the site laboratory ULN (upper limit of normal)
  * Hemoglobin less than 10.0 g/dL
  * Platelet count less than 100,000/mm3
  * Serum phosphate level below site laboratory LLN (lower limit of normal)
  * INR or aPTT greater than site laboratory ULN
  * Other safety tests (bicarbonate (HCO3), potassium (K), chloride (Cl), sodium (Na), calcium (Ca), fasting glucose) with results outside of the laboratories reference range
  * 1+ or greater protein on urine dipstick testing
  * 1+ or greater glucose on urine dipstick testing
* Culture-confirmed urinary tract infection
* Co-enrollment in any other HIV interventional research study (excluding behavioral only interventions) or prior enrollment in the active arm of a HIV vaccine trial.
* Clinically apparent or patient report of active skin disorders including: rash, pruritus, maculopapular rash, urticaria, vesiculobullous rash, and pustular rash.
* Women who are pregnant or breastfeeding.
* One or more reactive HIV rapid test results at screening or enrollment, even if HIV infection is not confirmed.
* Positive hepatitis B surface antigen (HBsAg) test.
* Excessive use of alcohol (more than 4 drinks a day on a regular basis).
* Interleukin therapy; medications with significant nephrotoxic potential, including but not limited to amphotericin B, aminoglycosides, cidofovir, foscarnet and systemic chemotherapy; and medications that may inhibit or compete for elimination via active renal tubular secretion (including but not limited to probenecid).
* Participants with a history of having a gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract or drug absorption.
* Intensive sampling cohort only:

  * A positive test for syphilis, gonorrhea, or Chlamydia
  * A positive test for HSV-2 (individuals with active lesions only)
  * Findings consistent with bacterial vaginosis, vaginal candidiasis, or trichomonas (women only)
  * History of STI within 3 months prior to enrollment
  * Medications that prolong clotting time (e.g., warfarin, heparin, clopidogrel classes.)
  * Abnormalities of the colorectal mucosa, or significant colorectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids).
  * Clinically apparent pelvic exam finding (observed by study staff) of genital lesions, erythema, edema or any other abnormal physical or pelvic exam finding that, in the opinion of the investigator or designee, would contraindicate study participation.
  * Women who have had cervical procedures (conization, LEEP procedure, cryosurgery) within the previous 6 months.
  * Spermicide as a method for contraception within last 30 days
* Any other reason or condition that in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Assess dose-proportionality | 49 days
  Assess dose-proportionality of intracellular TFV-DP and FTC-TP from weekly to daily dosing (Arms 1-4).
Comparison of intra-individual variability--days 28 and 35 | Days 28 and 35
  Describe intra-individual variability in intracellular TFV-DP and FTC-TP concentrations at steady-state (comparison of Day 28 and Day 35).

SECONDARY OUTCOMES:
Determine relationship between pre-dose and decaying concentrations | Days 35 and 49
  Describe the relationship between pre-dose and decaying concentrations of TFV, FTC, and their phosphorylated derivatives (TFV-DP and FTC-TP) in blood serum, peripheral blood mononuclear cells (PBMCs), CD4+ blood cells, total tissue cells, CD4+ tissue cells, tissue homogenate, semen, and luminal fluid at steady-state (Day 35 [pre-dose] and Day 49 [decaying, greater than one half-life for TFV-DP]).
Determine differences between men and women | 49 days
  Describe differences in intracellular TFV-DP and FTC-TP steady-state between men and women.
Safety profiles | 49 days
  Characterize the safety profiles of four different TDF/FTC PrEP regimens

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Study Chair — Johns Hopkins University; Kristine Patterson, MD, Study Chair — University of North Carolina; Kenneth Mayer, MD, Study Chair — Brown University; Adriana Andrade, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2010-11-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT01276600/Prot_ICF_000.pdf